CLINICAL TRIAL: NCT04163315
Title: Multimodal Connectome Study of Brain Tumor-operated Patients
Acronym: ConnecTC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-AOIP-01
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Brain
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dMRI, fMRI and electrocorticography (Experimental): With this exploratory pilot study, the investigator propose a multimodal evaluation of the structural and functional connectivity of patients with brain tumours, in order to better understand the tumor-induced lesion mechanisms on brain connectivity as well as the brain plasticity mechanisms that the brain develops to maintain a level of overall function neurological. The investigator hope to obtain multimodal brain mapping of locally brain-damaged patients, with a view to improving onco-functional neurosurgical practices.
  Interventions: Other: dMRI, fMRI and electrocorticography

INTERVENTIONS:
Other: dMRI, fMRI and electrocorticography — Patients included in the study will perform the pre-operative MRI (fMRI and fMRI) with a specific High Resolution Angular Diffusion (HARDI) sequence and a functional rest sequence. The additional scan time for this specific sequence is approximately 25 minutes, with no foreseeable negative impact on the patient

SUMMARY:
In this pilot study, the investigators propose a multimodal evaluation of the brain connectivity of brain tumor patients, in order to better understand the effects induced by focal lesions on brain structure and function, as well as brain plasticity mechanisms that may occur in such condition. The investigators aim at drawing a multimodal brain connectivity map of focally brain-damaged patients, with a view to improve onco-functional neurosurgical practices.

DETAILED DESCRIPTION:
Patients included in the present study will first perform the pre-operative MRI (dMRI and fMRI) with a specific High Resolution Angular Diffusion (HARDI) sequence and a functional acquisition at rest. Then, the investigators will record their cortico-cortical evoked potentials elicited by direct electrostimulation during the surgery, just before the tumor removal, following our usual protocol. Finally, all data (clinical, diffusion, electrical and functional connectivity) will be processed and correlated to each other.

ELIGIBILITY:
Inclusion Criteria:

* All patients with brain tumor for removal
* Age > 18 years
* Informed patient consent
* Membership of social security scheme

Exclusion Criteria:

* Contraindication to MRI
* Any subject with vascular stent implanted less than 6 weeks prior to the exam;
* Any subject carrying an intraocular or intracranial ferromagnetic foreign object close to nerve structures;
* Any subject carrying biomedical equipment such as a cardiac, neuronal or sensory pacemaker (cochlear implant) or a ventricular bypass valve without medical and paramedical supervision trained in the performance of MRI in these subjects;
* Presence of more than one brain tumor
* Refusal of patient participation
* Pregnant or nursing women. A urinary pregnancy test will be conducted for women of childbearing age. The results will be communicated to the patient by a doctor of her choice.
* Person staying in a health or social establishment
* Person in emergency situation
* Vulnerable patient: deprived of liberty, guardianship, curators, or safeguarding of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Correlations between tumor topography, cortical electrical conduction rates measured in electrocorticography, and microstructural measurements of white substance from diffusion MRI | 1 month

SECONDARY OUTCOMES:
Correlations between neurological disorders, tumor topography and network disruption identified in functional rest MRI | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ALMAIRAC, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, CHU de NICE, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sporns O. The human connectome: origins and challenges. Neuroimage. 2013 Oct 15;80:53-61. doi: 10.1016/j.neuroimage.2013.03.023. Epub 2013 Mar 23. PMID 23528922
- [Background] Duffau H. Stimulation mapping of white matter tracts to study brain functional connectivity. Nat Rev Neurol. 2015 May;11(5):255-65. doi: 10.1038/nrneurol.2015.51. Epub 2015 Apr 7. PMID 25848923
- [Background] Yeo BT, Krienen FM, Chee MW, Buckner RL. Estimates of segregation and overlap of functional connectivity networks in the human cerebral cortex. Neuroimage. 2014 Mar;88:212-27. doi: 10.1016/j.neuroimage.2013.10.046. Epub 2013 Nov 1. PMID 24185018
- [Background] Matsumoto R, Nair DR, LaPresto E, Najm I, Bingaman W, Shibasaki H, Luders HO. Functional connectivity in the human language system: a cortico-cortical evoked potential study. Brain. 2004 Oct;127(Pt 10):2316-30. doi: 10.1093/brain/awh246. Epub 2004 Jul 21. PMID 15269116